CLINICAL TRIAL: NCT01367795
Title: Surgical Procedures for Advanced Tumor Disease. A Prospective Study Evaluating Quality of Life
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Kantonsspital Olten (Other)
Responsible Party: Sponsor
Other Study IDs: EK 10/10; EK 2011/070 (Other: Ethikkommission Aargau/ Solothurn)
Record Dates: First submitted 2010-07-14; First posted 2011-06-07 (Estimated); Last update posted 2015-03-27 (Estimated); Status verified 2015-03

CONDITIONS: Advanced Cancer
Keywords: palliation; quality of life; surgery; surgery; palliative; lifestyle

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- palliative tumor disease: Patients in a known palliative setting with symptoms due to tumor growth.

SUMMARY:
Patients in a known palliative setting and with localized symptoms due to tumor growth will be evaluated for their quality of life before and after a surgical intervention (primary endpoint). Medical outcome in terms of length of stay in hospital, length of stay on a intensive care unit, complications, reinterventions will be recorded (secondary endpoints). The investigators will also observe patients with conservative treatment.

DETAILED DESCRIPTION:
What is the impact on quality of life by operations in symptomatic advanced tumor disease ? After informed consent patients in known palliative situations and with localized symptoms due to tumor growth will be enrolled in our study. The investigators will assess Quality of life with the EORTC QLQ C30-questionnaire and collect data about the disease an the actual state of the patients.

By the time of discharge out of hospital the investigators will hand out the questionnaire again and the investigators will collect data regarding the therapies, operations, complications, reinterventions, time spent on a intensive care unit, time spent in hospital.

The questionnaire will be completed after 4 and 12 weeks as well.

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* tumor patients within a known palliative situation, patients do know about the absence of a curative treatment
* patients are symptomatic because of localized tumor growth
* patients having an operation for symptom relief or treated without surgery

Exclusion Criteria:

* patients with an only intraoperatively seen palliative tumor disease
* debulking operations, prophylactic operations for prevention of symptoms, operations for venous access (an exception will be made for enteric bypass operations in patients with a yet preserved passage)
* dementia, age ≤ 18, barrier of speech

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in a known tumorrelated palliative situation will be included when an operation is discussed for relieve of symptomatic localised tumor growth . Patients will be recruited from clinics or the emergency room.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2010-07; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Quality of life 4 weeks after palliative surgery | 4 weeks after palliative surgery
  Quality of life will be measured by the questionnaire EORTC-QLQ-C30 (European Organization for Research and Treatment of Cancer-Quality of Life).

SECONDARY OUTCOMES:
duration of stay in hospital | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks
duration of stay in an intensive care unit | participants will be followed for the duration of stay in an intensive care unit, an expected average of 0 to 2 days
complications | the participants will be followed for the duration of hospital stay, an expected average of 2 weeks
  Complications will be recorded following the Clavien-Dindo classification of surgical complications. This 5-scale classification is based on the type of therapy needed to correct the complications.
reoperations | the participants will be followed for the duration of hospital stay, an expected average of 2 weeks
  The need for reoperations is generally part of the 5-class complication scale by Clavien and Dindo, which we are using to record complications. Reoperations (class IIIb in the classification of complications) are recorded seperately.

CONTACTS AND LOCATIONS:
Overall Officials: Carsten T. Viehl, MD, Principal Investigator — Department of Surgery, University Hospital of Basel
Locations (2):
- Switzerland (2):
  - Hospital Biel, Department for Surgery, Basel, Basel
  - Kantonsspital Olten, Department for Surgery, Olten, Canton of Solothurn